CLINICAL TRIAL: NCT05373511
Title: Evaluation of Body Posture and Postural Balance Among Young Adults With Bronchial Asthma in the United Arab Emirates - A Correlational Cross Sectional Study
Brief Title: Assessing Body Posture and Postural Balance Among Young Adults With Bronchial Asthma
Status: Completed | Type: Observational
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Other Study IDs: REC-22-01-12
Record Dates: First submitted 2022-04-15; First posted 2022-05-13 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-10

CONDITIONS: Bronchial Asthma
Keywords: body Posture; dynamic Balance; Biodex Balance System; DIERS FORMETRIC 4D posture analysis
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bronchial asthma: Inclusion criteria:
  Participants over the age of 18 who have had mild to moderate bronchial asthma since childhood and have been referred by a pulmonologist or physician
  Exclusion criteria:
  Participants with other health issues such as cardiorespiratory issues, neurological deficits or diseases such as nerve compressions, any chronic diseases or suffering from respiratory tract infections, participants with a history of previous serious injuries to the musculoskeletal system, which may result in body posture disturbances Any disease that impairs one's sense of balance
  Interventions: Other: 3D/4D spine and posture analysis "DIERS FORMETRIC 4D" ,The Biodex Balance System SD-
- non-asthmatic control group:: Inclusion and Exclusion criteria for non-asthmatic control group:
  Inclusion criteria:
  For the healthy subjects referred by a consultant pulmonologist/physician, age- and gender-matched volunteers were recruited from the community
  Exclusion criteria:
  Other health issues, such as cardiorespiratory issues, neurological deficits, musculoskeletal problems, and peripheral vascular diseases& pregnancy may affect test performance.
  Interventions: Other: 3D/4D spine and posture analysis "DIERS FORMETRIC 4D" ,The Biodex Balance System SD-

INTERVENTIONS:
Other: 3D/4D spine and posture analysis "DIERS FORMETRIC 4D" ,The Biodex Balance System SD- — 3D/4D spine and posture analysis "DIERS FORMETRIC 4D" for postural analysis assessment
  ,The Biodex Balance System SD- for balance assessment

SUMMARY:
The purpose of the study is to assess the relationship between body posture and dynamic balance in adults with childhood-onset asthma and compare them to a non-asthmatic control group matched for gender, age, weight, and height.

DETAILED DESCRIPTION:
Participants will sign a consent form and provide personal information such as gender, age, weight, and height for calculating BMI, pulmonary function test, and respiratory muscle strength test, as well as their asthmatic/clinical history. After collecting demographic information and obtaining consent from participants, they will be asked to remove their T-shirts and stand in the usual relaxed standing position facing the opposite side of the machine's window. When the machine is properly positioned, it will take photographs. which will then be converted into three-dimensional images on the computer for further analysis. When the participant is fully dressed and ready, the second test will be performed using the Biodex balance machine. The parameters and testing mode to begin the dynamic balance test will be entered into the machine, and the procedure will begin. The participants will be thanked for their participation and contribution to our study

ELIGIBILITY:
Inclusion Criteria:

* For the healthy subjects referred by a consultant pulmonologist/physician
* age- and gender-matched volunteers were recruited from the community

Exclusion Criteria:

* Other health issues, such as cardiorespiratory issues, neurological deficits
* musculoskeletal problems and peripheral vascular diseases& pregnancy may affect test performance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: bronchial asthma -18 years above health group ( non bronchial asthma )
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
body posture assessment using DIERS FORMETRIC 4D, | baseline
  From a single image, the instrument will generate 40 named spine shape parameters, like( lateral deviation (mm), trunk imbalance (mm), shoulder tilt (mm) )
postural balance assessment by biodex balance system machine | baseline
  Double Leg Eyes Open (DLEO) Degree (angle), Double Leg Eyes Closed (DLEC) Degree (angle), Single Leg Eyes Open (SLEO) Degree (angle), single Leg Eyes closed (SLEC) Degree (angle), Overall Balance/stability Index (OBI/OSI )Degree (angle), ANT/POST Balance Index (APBI )Degree (angle), MED/LAT Balance Index (MLBI)Degree (angle),

CONTACTS AND LOCATIONS:
Overall Officials: Arthur De Sa Ferreira, phd, Study Chair — Augusto Motta University Centre
Locations (1):
- Gopala Krishna Alaparthi, Sharjah city, UAE, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: very month
Access Criteria: through mail

REFERENCES:
- [Derived] Alaparthi GK, Moustafa IM, Lopes AJ, Ferreira AS. Pulmonary function, body posture and balance in young adults with asthma: A cross-sectional study. PLoS One. 2025 Mar 3;20(3):e0316663. doi: 10.1371/journal.pone.0316663. eCollection 2025. PMID 40029906